CLINICAL TRIAL: NCT00157729
Title: Evaluation of the Effects of MC-1 Alone and in Combination With an ACE Inhibitor on Ambulatory Blood Pressure and Metabolic Function in Hypertensive Patients With Type 2 Diabetes Mellitus
Brief Title: MATCHED (MC-1 and ACE Therapeutic Combination for Hypertensive Diabetics)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicure (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MC6021-CL-04001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-10-31 (Estimated); Status verified 2006-10

CONDITIONS: Diabetes Mellitus Type 2; Hypertension; Metabolic Syndrome
Keywords: Hypertension; antihypertensive agents; diabetes mellitus type 2; metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Metabolic Syndrome | interventions — Pyridoxal Phosphate; Angiotensin-Converting Enzyme Inhibitors

INTERVENTIONS:
Drug: pyridoxal-5'-phosphate with and without ACE inhibitor

SUMMARY:
The purpose of this study is to determine whether MC-1 alone and in combination with an ACE inhibitor is effective in reducing blood pressure and metabolic dysfunctions associated with diabetes

DETAILED DESCRIPTION:
Hypertension is an extremely common co-morbid condition in diabetics, affecting up to 11 million patients, depending on obesity, ethnicity and age. Hypertension substantially increases the risk of both macrovascular and microvascular complications including stroke, coronary artery disease, peripheral vascular disease, retinopathy, nephropathy and possibly neuropathy.

In recent years, adequate data from well-designed randomized clinical trials have demonstrated the effectiveness of aggressive treatment of hypertension in reducing diabetic complications. In the epidemiological UK Prospective Diabetes Study (UKPDS), each 10 mmHg decrease in mean systolic blood pressure was associated with reductions in risk of 12% for any complication related to diabetes, 15% for deaths related to diabetes, 11% for myocardial infarction and 13% for microvascular complications. Currently the consensus guidelines recommend a blood pressure target of <130/80 mmHg in diabetic patients with hypertension, even though they recognize many people will require three or more drugs to reach this goal.

MC-1 is a naturally occurring metabolite of vitamin B6, and thus has very low toxicity. Evidence from pre-clinical studies suggests that MC-1 has beneficial effects on hypertension and metabolic dysfunction. This trial will assess the effects of MC-1 alone and MC-1 in combination with an ACE inhibitor compared to placebo on hypertension and parameters of metabolic function in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus treated with diet, oral hypoglycaemic agents or insulin) for a minimum of 2 years (24 months)
* Systolic hypertension prior to entry into the washout period. At Visit 3 patients must have a mean sitting systolic blood pressure in the range of 140-180 mmHg, and a mean sitting diastolic blood pressure <110mmHg
* A mean daytime ambulatory systolic blood pressure greater than or equal to 135 mm Hg at baseline

Exclusion Criteria:

* Poorly controlled type 2 diabetes mellitus (HbA1c ≥ 10%)
* Secondary hypertension of any aetiology, such as renal artery stenosis, coarctation of the aorta or pheochromocytoma
* History of malignant hypertension
* Body mass index > 37
* Single functioning kidney
* Known sensitivity or intolerance to angiotensin-converting enzyme inhibitors
* History of angioedema
* Known syncopal disorder
* Pregnant woman or a woman of childbearing potential who is sexually active and not using an appropriate method of birth control (double barrier or oral contraceptives)
* Concomitant therapy with any antihypertensive medications, including those used for indications other than hypertension (e.g., diuretics for any reason, minoxidil for hair loss, propranolol HCl for migraine, terazosin HCl for benign prostatic hyperplasia, 5-phosphodiesterase inhibitors (Viagra, Cialis, Levitra) within 48 hours of clinic visit, ACE-inhibitors for congestive heart failure, or any agent which could cause a change in blood pressure), except for stable doses of NSAIDs, or tricyclic agents taken at bedtime. Patients who are unwilling to discontinue these medications or patients in whom the Investigator feels it is clinically inappropriate to discontinue these medications should not participate in the study
* Concomitant therapy with lithium and/or major psychotropic agents such as phenothiazines
* Concomitant therapy with oral steroids or ACTH
* Concomitant therapy with cold and/or flu medications containing sympathomimetic agents. Intermittent use of therapies containing ephedrine is permitted except within 72 hours of clinic visits for mean trough SiSBP
* Concomitant therapy with any vitamin supplement that may contain pyridoxine or pyridoxine derivative such as pyridoxal phosphate or pyridoxal
* Hypertension induced by oral contraceptives. Replacement hormones (thyroid, testosterone, estrogens) are permitted if the patient has been on a stable dose for at least three months
* Existing symptomatic cerebro-vascular disease including previous transient ischemic attack (TIA) or stroke within 12 months prior to screening
* Myocardial infarction, percutaneous coronary intervention and coronary artery bypass surgery within 6 months prior to screening
* Clinically significant AV conduction disturbance, i.e., second or third degree AV block, sick sinus syndrome or clinically significant bradycardia (resting heart rate < 60 beats/minute) without a permanent pacemaker
* Presence of atrial flutter or atrial fibrillation
* Potentially life-threatening ventricular arrhythmias, decompensated valvular disease, presence of hemodynamically significant obstructive valvular disease, or cardiomyopathy
* Serum potassium < 3.5 or > 5.5 mEq/L
* The presence of severe hepatic impairment as manifested by AST (SGOT) > 2.5 times the upper limit of normal or ALT (SGPT) > 2.5 times the upper limit of normal
* Any clinically significant laboratory value which in the Investigator's judgement could be clinically significant to the outcome of this study. This includes, but is not limited to, hematocrit, haemoglobin or platelet count
* Any moderate to severe renal impairment, as manifested by serum creatinine more than 200 micromol/L
* A history of clinically important gastrointestinal resection, malabsorption or cirrhosis of the liver
* Any concurrent severe disease that, in the Investigator's judgement, could preclude participation or survival
* Use of any investigational drug or device, or participation in any drug study during or within 30 days prior to baseline
* Inability to be taken off of all current antihypertensive medications
* Unwillingness or inability to give consent or to follow the protocol procedures
* Arm circumference greater than 41 cm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
Effects on blood pressure:
Determine the efficacy of MC-1 and of the combination of MC-1/ACE inhibitor on blood pressure as measured by mean daytime ambulatory systolic blood pressure.
Effects on metabolic function:
Determine the efficacy of MC-1 and of the combination of MC-1/ACE inhibitor on metabolic function as measured by insulinemia, fasting serum glucose, glycated hemoglobin, and triglycerides.

SECONDARY OUTCOMES:
To compare the effects of the different treatment regimens as measured by:
mean change from baseline in mean daytime ambulatory diastolic BP
mean change from baseline in mean 24 hour and mean night-time ambulatory systolic BP
mean changes from baseline in mean 24 hour, mean daytime and mean night-time pulse pressure
mean changes from baseline in clinic trough sitting systolic BP (SiSBP)
mean changes from baseline in mean 24 hour, and mean night-time ambulatory diastolic BP
mean changes from baseline in clinic trough sitting diastolic BP (SiDBP)
mean change in endothelial function as measured by mean changes in different markers such as ICAM-1, VCAM-1, E-selectin and albuminuria
mean changes in C-reactive protein (CRP)
mean changes in homocysteine
mean changes in creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Yves Lacourciere, MD, FRCP, Principal Investigator — Centre Hospitalier de l'Universite Laval
Locations (1):
- Centre Hospitalier Université Laval, Sainte-Foy, Quebec, Canada